CLINICAL TRIAL: NCT02683317
Title: Effect of Enteral Administration of Docosahexaenoic Acid on Development of the Retinopathy of Prematurity
Brief Title: Enteral Administration of Docosahexaenoic Acid to Prevent Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mariela Bernabe García, Full Time Researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R-2015-785-051
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Retinopathy of Prematurity
Keywords: DHA; Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Docosahexaenoic Acids; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Regarding the Study phase, the intervention was a nutraceutical, docosahexaenoic acid, derived from omega 3 fatty acid family.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA group (Experimental): Experimental group will receive 75 mg of docosahexaenoic acid per kilo of baseline weight in one dose per day, administered by enteral feeding throughout 14 days.
  Interventions: Dietary Supplement: docosahexaenoic acid
- Control group (Sham Comparator): Control group will receive sunflower oil, the excipient of the DHA in our intervention.
  They will receive it once a day, administered by enteral feeding throughout 14 days.
  Interventions: Dietary Supplement: sunflower oil

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid — Docosahexaenoic acid is a dietary supplement derived from algae.
  Other Names: n-3 long chain polyunsaturated fatty acid
  Arms: DHA group
Dietary Supplement: sunflower oil — Sunflower similar to the excipient used in experimental group
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate whether docosahexaenoic acid given by enteral feeding prevent retinopathy of prematurity and/or diminish its severity in preterm infants.

DETAILED DESCRIPTION:
Preterm neonates who start receiving enteral feeding will receive the intervention with docosahexaenoic acid (DHA) since the first day and throughout 14 days, one dose per day.

The opthalmic evaluation will be done after 4-5 weeks after birth and followed until 42-45 corrected gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 g
* Plan to feed by enteral way at a short term
* Written informed consent, signed by both parents.

Exclusion Criteria:

* Congenital malformations that avoid enteral feeding
* immunosuppressor diseases
* Need for major surgery
* Persistent bleeding at any level
* Mother taking n-3 supplements and planning to breastfed
* Parents who decline the authorization for participating in the study
* Early discharge to other hospital outside the metropolitan area

Ages: 60 Minutes to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Presence of retinopathy of prematurity (ROP) | ROP will be evaluated from 4 to 5 weeks after birth throughout 42-45 of corrected gestational age.
  The medical screening to determine the presence ROP will include the exhaustive search of injury on the zone, stage and the presence of plus disease in retina of the preterm infants. The measure unit is frequency of ROP (presence =1 or absence=0) registering the corrected gestational age of the first identification.

SECONDARY OUTCOMES:
Severity of ROP | ROP will be evaluated as changes in each retina's eye from 4 to 5 weeks after birth throughout 42-45 of corrected gestational age
  The study will determine the severity of retinopathy of prematurity as ordinal variable with frequencies, according to the following classification:
  1. ROP stage 1 or threshold needs treatment:
     * ROP in Zone I any stage if it is associate to presence of Plus.
     * ROP stage 1 in Zone I + Plus disease
     * ROP stage 2 in Zone I + Plus disease
     * ROP stage 3 in Zone I + Plus disease
     * ROP in Zone I Stage 3 with or without Plus disease.
     * ROP in Zone II Stage 2 or 3 + Plus disease.
  2. ROP Stage 2 or pre-threshold, require close monitoring:
     * ROP in Zone I, Stage 1 or 2 without Plus
     * ROP in Zone II, Stage 3 without Plus
  3. ROP in zone II or III, Stage 1 or 2 without Plus, require periodic monitoring.
  4. ROP in remission
  5. Without retinopathy

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Bernabe-Garcia, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Research in Nutrition, Pediatric Hospital, Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, Del Prado M, Rivera D, Ruiz G, Maldonado J, Villegas R. Docosahexaenoic acid administered in the acute phase protects the nutritional status of septic neonates. Nutrition. 2006 Jul-Aug;22(7-8):731-7. doi: 10.1016/j.nut.2006.04.002. Epub 2006 Jun 5. PMID 16750345
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, del Valle O, Gonzalez-Moreno G, Martinez-Basilea A, Villegas R. Oral administration of docosahexaenoic acid attenuates interleukin-1beta response and clinical course of septic neonates. Nutrition. 2012 Apr;28(4):384-90. doi: 10.1016/j.nut.2011.07.016. Epub 2011 Nov 12. PMID 22079797
- [Background] Bernabe-Garcia M, Lopez-Alarcon M, Villegas-Silva R, Mancilla-Ramirez J, Rodriguez-Cruz M, Maldonado-Hernandez J, Chavez-Rueda KA, Blanco-Favela F, Espinoza-Garcia L, Lagunes-Salazar S. Beneficial Effects of Enteral Docosahexaenoic Acid on the Markers of Inflammation and Clinical Outcomes of Neonates Undergoing Cardiovascular Surgery: An Intervention Study. Ann Nutr Metab. 2016;69(1):15-23. doi: 10.1159/000447498. Epub 2016 Jul 9. PMID 27394149
- [Background] Bernabe-Garcia M, Lopez-Alarcon M, Salgado-Sosa A, Villegas-Silva R, Maldonado-Hernandez J, Rodriguez-Cruz M, Rivas-Ruiz R, Chavez-Sanchez L, Blanco-Favela FA, Mancilla-Ramirez J, Gordillo-Alvarez V, Madrigal-Muniz O. Enteral Docosahexaenoic Acid Reduces Analgesic Administration in Neonates Undergoing Cardiovascular Surgery. Ann Nutr Metab. 2016;69(2):150-160. doi: 10.1159/000452227. Epub 2016 Nov 2. PMID 27806350
- [Result] Bernabe-Garcia M, Villegas-Silva R, Villavicencio-Torres A, Calder PC, Rodriguez-Cruz M, Maldonado-Hernandez J, Macias-Loaiza D, Lopez-Alarcon M, Inda-Icaza P, Cruz-Reynoso L. Enteral Docosahexaenoic Acid and Retinopathy of Prematurity: A Randomized Clinical Trial. JPEN J Parenter Enteral Nutr. 2019 Sep;43(7):874-882. doi: 10.1002/jpen.1497. Epub 2019 Jan 6. PMID 30614004